CLINICAL TRIAL: NCT04298034
Title: Randomized Controlled Trial for Postpartum Antihypertensive Treatment of Women With Preeclampsia
Brief Title: Preeclampsia Postpartum Antihypertensive Treatment
Acronym: P-PAT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO36760
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia; Hypertension in Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Labetalol; Nifedipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician will be masked to which group the patient was randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): The patients randomized to the treatment group will have an antihypertensive medication prescribed to them. The specific medication will be either labetalol or nifedipine based on allergies and clinically appropriateness of the medication. The patient will be instructed on the dosing, timing, and possible adverse effects.
  Interventions: Drug: Labetalol, Nifedipine
- No-treatment (No Intervention)

INTERVENTIONS:
Drug: Labetalol, Nifedipine — Antihypertensive treatment that is safe and well studied in peripartum women.
  Other Names: Procardia; Trandate, Normodyne
  Arms: Treatment

SUMMARY:
The goal of this study is to compare whether antihypertensive treatment in the postpartum period decreases postpartum hypertension and its associated maternal morbidity, including risk of readmission and healthcare utilization in comparison with no treatment. Women with preeclampsia diagnosed during the antepartum, intrapartum or postpartum period will be randomized to either initiate antihypertensive treatment or standard of care. We hypothesize that postpartum antihypertensive treatment of patients with preeclampsia will decrease risk of hospital readmission, healthcare utilization and the number of severe range blood pressures at postpartum follow-up visits.

DETAILED DESCRIPTION:
This will be a randomized, controlled trial of 300 women with a diagnosis of preeclampsia at any point in their current pregnancy or immediately postpartum. Immediately postpartum is defined as preeclampsia diagnosed after delivery but prior to discharge from the hospital. The diagnosis of preeclampsia will be made using standardized definitions by the American College of Obstetrics and Gynecology. Preeclampsia is diagnosed with new-onset hypertension of blood pressure of greater than or equal to 140 systolic blood pressure or greater than or equal to 90 diastolic blood pressure recorded twice at least four hours apart AND proteinuria, defined as 300mg of protein in a 24hour urine collection or a protein/creatinine ratio of 0.3. If the above blood pressure criteria are met and there is not proteinuria, preeclampsia can still be diagnosed if there is thrombocytopenia with platelet count of less than 100,000, renal insufficiency with creatinine of greater than 1.1 or twice the patient's individual baseline, impaired liver function with AST or ALT twice normal or epigastric/right upper quadrant pain, pulmonary edema, new-onset headache unresponsive to medication, or visual disturbance. All of these findings should not be explained by an alternative diagnosis.

Women will be consented and randomized at the time of their diagnosis, within 96 hours of their delivery. The patients randomized to the treatment group will have an antihypertensive medication prescribed to them. The specific medication will be either labetalol, nifedipine or hydralazine based on allergies and clinically appropriateness of the medication. The patient will be instructed on the dosing, timing, and possible adverse effects. All subject's blood pressures will be monitored per standard postpartum protocols. As per standard practice, all patients with preeclampsia will be asked to return at 7-10 days for a blood pressure check and then again at 6 weeks for a complete postpartum assessment.

Consent of patients, review of blood pressures, data collection and storage, and statistical analysis will be performed at the Medical College of Wisconsin (MCW) through the Maternal Fetal medicine department. Women will be allowed to continue routine antenatal, intrapartum and postpartum care with their primary obstetrician. The research team will follow enrolled patients through the 6-week postpartum follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Immediately postpartum (delivered in previous 96 hours)
* Diagnosed with preeclampsia during pregnancy, labor or immediately postpartum
* >30% of blood pressures in the postpartum period were elevated (systolic 140 or higher OR diastolic 90 or higher)

Exclusion Criteria:

* Chronic hypertension with superimposed preeclampsia
* Diagnosis of preeclampsia after discharge from delivery hospitalization
* Persistent severe range blood pressures after delivery requiring initiation of antihypertensive regimen by the care team
* >50% of blood pressures in the postpartum period were normal (systolic less than 140 AND diastolic less than 90)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission | Within 6 weeks from delivery

SECONDARY OUTCOMES:
Rate of Healthcare Utilization | Within 6 weeks from delivery
  hospital readmissions, increased number of postpartum visits or phone calls, emergency room or urgent care visits, consultation with primary care (internal medicine, family medicine), cardiology, or maternal-fetal-medicine specialists
percentage of severe range blood pressures at the 7-10 days postpartum visit | 7-10 days postpartum
percentage of severe range blood pressures at the 6 week postpartum visit | Approximately 6 weeks postpartum
compare mean systolic and mean diastolic blood pressure values at 7-10 days postpartum and at 6weeks postpartum | 6 weeks pospartum

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin-Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sibai BM. Hypertensive disorders of pregnancy: the United States perspective. Curr Opin Obstet Gynecol. 2008 Apr;20(2):102-6. doi: 10.1097/GCO.0b013e3282f73380. No abstract available. PMID 18388806
- [Background] Mogos MF, Salemi JL, Spooner KK, McFarlin BL, Salihu HH. Hypertensive disorders of pregnancy and postpartum readmission in the United States: national surveillance of the revolving door. J Hypertens. 2018 Mar;36(3):608-618. doi: 10.1097/HJH.0000000000001594. PMID 29045342
- [Background] Tan LK, de Swiet M. The management of postpartum hypertension. BJOG. 2002 Jul;109(7):733-6. doi: 10.1111/j.1471-0528.2002.01012.x. No abstract available. PMID 12135206
- [Background] Ade-Conde JA, Alabi O, Higgins S, Visvalingam G. Maternal post natal hospital readmission-trends and association with mode of delivery. Ir Med J. 2011 Jan;104(1):17-20. PMID 21387880
- [Background] Clapp MA, Little SE, Zheng J, Robinson JN. A multi-state analysis of postpartum readmissions in the United States. Am J Obstet Gynecol. 2016 Jul;215(1):113.e1-113.e10. doi: 10.1016/j.ajog.2016.01.174. PMID 27829570
- [Background] Ferrazzani S, De Carolis S, Pomini F, Testa AC, Mastromarino C, Caruso A. The duration of hypertension in the puerperium of preeclamptic women: relationship with renal impairment and week of delivery. Am J Obstet Gynecol. 1994 Aug;171(2):506-12. doi: 10.1016/0002-9378(94)90290-9. PMID 8059832
- [Background] Kassebaum NJ, Bertozzi-Villa A, Coggeshall MS, Shackelford KA, Steiner C, Heuton KR, Gonzalez-Medina D, Barber R, Huynh C, Dicker D, Templin T, Wolock TM, Ozgoren AA, Abd-Allah F, Abera SF, Abubakar I, Achoki T, Adelekan A, Ademi Z, Adou AK, Adsuar JC, Agardh EE, Akena D, Alasfoor D, Alemu ZA, Alfonso-Cristancho R, Alhabib S, Ali R, Al Kahbouri MJ, Alla F, Allen PJ, AlMazroa MA, Alsharif U, Alvarez E, Alvis-Guzman N, Amankwaa AA, Amare AT, Amini H, Ammar W, Antonio CA, Anwari P, Arnlov J, Arsenijevic VS, Artaman A, Asad MM, Asghar RJ, Assadi R, Atkins LS, Badawi A, Balakrishnan K, Basu A, Basu S, Beardsley J, Bedi N, Bekele T, Bell ML, Bernabe E, Beyene TJ, Bhutta Z, Bin Abdulhak A, Blore JD, Basara BB, Bose D, Breitborde N, Cardenas R, Castaneda-Orjuela CA, Castro RE, Catala-Lopez F, Cavlin A, Chang JC, Che X, Christophi CA, Chugh SS, Cirillo M, Colquhoun SM, Cooper LT, Cooper C, da Costa Leite I, Dandona L, Dandona R, Davis A, Dayama A, Degenhardt L, De Leo D, del Pozo-Cruz B, Deribe K, Dessalegn M, deVeber GA, Dharmaratne SD, Dilmen U, Ding EL, Dorrington RE, Driscoll TR, Ermakov SP, Esteghamati A, Faraon EJ, Farzadfar F, Felicio MM, Fereshtehnejad SM, de Lima GM, Forouzanfar MH, Franca EB, Gaffikin L, Gambashidze K, Gankpe FG, Garcia AC, Geleijnse JM, Gibney KB, Giroud M, Glaser EL, Goginashvili K, Gona P, Gonzalez-Castell D, Goto A, Gouda HN, Gugnani HC, Gupta R, Gupta R, Hafezi-Nejad N, Hamadeh RR, Hammami M, Hankey GJ, Harb HL, Havmoeller R, Hay SI, Pi IB, Hoek HW, Hosgood HD, Hoy DG, Husseini A, Idrisov BT, Innos K, Inoue M, Jacobsen KH, Jahangir E, Jee SH, Jensen PN, Jha V, Jiang G, Jonas JB, Juel K, Kabagambe EK, Kan H, Karam NE, Karch A, Karema CK, Kaul A, Kawakami N, Kazanjan K, Kazi DS, Kemp AH, Kengne AP, Kereselidze M, Khader YS, Khalifa SE, Khan EA, Khang YH, Knibbs L, Kokubo Y, Kosen S, Defo BK, Kulkarni C, Kulkarni VS, Kumar GA, Kumar K, Kumar RB, Kwan G, Lai T, Lalloo R, Lam H, Lansingh VC, Larsson A, Lee JT, Leigh J, Leinsalu M, Leung R, Li X, Li Y, Li Y, Liang J, Liang X, Lim SS, Lin HH, Lipshultz SE, Liu S, Liu Y, Lloyd BK, London SJ, Lotufo PA, Ma J, Ma S, Machado VM, Mainoo NK, Majdan M, Mapoma CC, Marcenes W, Marzan MB, Mason-Jones AJ, Mehndiratta MM, Mejia-Rodriguez F, Memish ZA, Mendoza W, Miller TR, Mills EJ, Mokdad AH, Mola GL, Monasta L, de la Cruz Monis J, Hernandez JC, Moore AR, Moradi-Lakeh M, Mori R, Mueller UO, Mukaigawara M, Naheed A, Naidoo KS, Nand D, Nangia V, Nash D, Nejjari C, Nelson RG, Neupane SP, Newton CR, Ng M, Nieuwenhuijsen MJ, Nisar MI, Nolte S, Norheim OF, Nyakarahuka L, Oh IH, Ohkubo T, Olusanya BO, Omer SB, Opio JN, Orisakwe OE, Pandian JD, Papachristou C, Park JH, Caicedo AJ, Patten SB, Paul VK, Pavlin BI, Pearce N, Pereira DM, Pesudovs K, Petzold M, Poenaru D, Polanczyk GV, Polinder S, Pope D, Pourmalek F, Qato D, Quistberg DA, Rafay A, Rahimi K, Rahimi-Movaghar V, ur Rahman S, Raju M, Rana SM, Refaat A, Ronfani L, Roy N, Pimienta TG, Sahraian MA, Salomon JA, Sampson U, Santos IS, Sawhney M, Sayinzoga F, Schneider IJ, Schumacher A, Schwebel DC, Seedat S, Sepanlou SG, Servan-Mori EE, Shakh-Nazarova M, Sheikhbahaei S, Shibuya K, Shin HH, Shiue I, Sigfusdottir ID, Silberberg DH, Silva AP, Singh JA, Skirbekk V, Sliwa K, Soshnikov SS, Sposato LA, Sreeramareddy CT, Stroumpoulis K, Sturua L, Sykes BL, Tabb KM, Talongwa RT, Tan F, Teixeira CM, Tenkorang EY, Terkawi AS, Thorne-Lyman AL, Tirschwell DL, Towbin JA, Tran BX, Tsilimbaris M, Uchendu US, Ukwaja KN, Undurraga EA, Uzun SB, Vallely AJ, van Gool CH, Vasankari TJ, Vavilala MS, Venketasubramanian N, Villalpando S, Violante FS, Vlassov VV, Vos T, Waller S, Wang H, Wang L, Wang X, Wang Y, Weichenthal S, Weiderpass E, Weintraub RG, Westerman R, Wilkinson JD, Woldeyohannes SM, Wong JQ, Wordofa MA, Xu G, Yang YC, Yano Y, Yentur GK, Yip P, Yonemoto N, Yoon SJ, Younis MZ, Yu C, Jin KY, El Sayed Zaki M, Zhao Y, Zheng Y, Zhou M, Zhu J, Zou XN, Lopez AD, Naghavi M, Murray CJ, Lozano R. Global, regional, and national levels and causes of maternal mortality during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Sep 13;384(9947):980-1004. doi: 10.1016/S0140-6736(14)60696-6. Epub 2014 May 2. PMID 24797575
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Levine LD, Nkonde-Price C, Limaye M, Srinivas SK. Factors associated with postpartum follow-up and persistent hypertension among women with severe preeclampsia. J Perinatol. 2016 Dec;36(12):1079-1082. doi: 10.1038/jp.2016.137. Epub 2016 Sep 1. PMID 27583396
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 203: Chronic Hypertension in Pregnancy. Obstet Gynecol. 2019 Jan;133(1):e26-e50. doi: 10.1097/AOG.0000000000003020. PMID 30575676
- [Background] Boffa RJ, Constanti M, Floyd CN, Wierzbicki AS; Guideline Committee. Hypertension in adults: summary of updated NICE guidance. BMJ. 2019 Oct 21;367:l5310. doi: 10.1136/bmj.l5310. No abstract available. PMID 31636059